CLINICAL TRIAL: NCT04879160
Title: Systematically Assessing Changes in Plexiform Neurofibroma Related Disfigurement From Photographs of Subjects With Neurofibromatosis Type 1 on a Phase 2 Clinical Trial
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10000173; 000173-C
Record Dates: First submitted 2021-05-07; First posted 2021-05-10 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Neurofibromatosis 1
Keywords: Selumetinib; novel disfigurement scale; Natural History
MeSH Terms: conditions — Neurofibromatosis 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 1/ Cohort 1A: Clinician raters familiar with NF1
- 2/ Cohort 1B: Clinician raters without specific NF1 familiarity
- 3/ Cohort 2A: Non-clinician raters familiar with NF1
- 4/ Cohort 2B: Non-clinician raters without specific NF1 familiarity
- 5/ Cohort 3: Subjects with NF1

SUMMARY:
Background:

People with Neurofibromatosis type 1 (NF1) have an increased risk of developing plexiform neurofibromas (PNs). PNs are tumors that form in the tissue. They can form anywhere in the body. They can become visible and cause deformations. Researchers want to see if selumetinib changes how PNs look in people with NF1. They also want to test a rating system for the visibility of these tumors.

Objective:

To see if treatment with selumetinib can improve the appearance of visible PNs in people with NF1, as determined by people who are/are not familiar with NF1.

Eligibility:

People with NF1 who have one or more visible PNs and have been enrolled in study 11C0161 or 08C0079. Clinicians and non-clinicians with and without experience in NF1 are also needed to serve as raters.

Design:

Participants are people with NF1 who had photos taken on study 11C0161 or 08C0079. Raters are people who will evaluate the PNs in the photos. They will rate the tumors on a scale from 1 to 10, from less to most visible.

Participants medical records will be reviewed. Their photos will be shown to 28 raters.

Raters will fill out a survey about their demographics, place of work, and if they are familiar with NF1. They will view sample photos to learn how PNs look and how to rate PNs.

Raters will view photos of PNs taken before and after selumetinib treatment. They will also view photos of PNs that were not treated. They will rate PNs for up to 40 participants. They will have 1-2 sessions. Each session will last 1 hour....

DETAILED DESCRIPTION:
Background:

Up to 50% of subjects with Neurofibromatosis Type 1 (NF1) will develop histologically benign plexiform neurofibromas (PN).

One of the most common morbidities associated with PN is a disfigurement that has the potential to pose formidable obstacles to the medical and psychosocial well-being of subjects with NF1.

The phase 2 trial of the MEK inhibitor selumetinib for inoperable PN (NCT01362803) have shown volumetric shrinkage of PN in approximately 74% of subjects with at least one PN morbidity, with most of the responsive tumors decreasing in size by 20-50% volume from baseline. Both trials have completed enrollment and primary study objectives.

In this selumetinib trial, standardized photography of visible PN was performed over time to assess for changes in disfigurement over time. This trial did not include criteria to measure changes in disfigurement and no validated criteria for measurement of PN-related disfigurement exist.

We developed a scale to rate the extent of a disfigurement from NF1 PN and will apply this scale to photographs obtained on the phase II selumetinib trial.

Objective:

To determine if selumetinib treatment is associated with improvement in PN-related disfigurement, as determined by raters reviewing photographs before treatment and just prior to cycle 13 of treatment.

Eligibility:

Four groups of adult raters to rate disfigurement who are not directly involved in the conduct of the selumetinib treatment study (NCT01362803), who are not NIH employees, and can read and write in English.

Design:

-Methods

Photographs of consenting individuals with PN, who may or may not have received selumetinib will be reviewed.

Raters will be presented pre and post treatment photographs of persons who received selumetinib as well as control photographs of persons not receiving selumetinib.

Each rater is presented with the same set of photographs though placement and order may differ.

Each rater will look at photographs of each individual with PN for at least 10 seconds, then with photos still visible, raters will verbally answer a questionnaire.

The rater will be asked questions at the end of the session to assess the feasibility of the questionnaire.

Session will be repeated by some raters approximately six months later on a subset of the photographs.

-Statistical Analysis

In each cohort of raters, for each subject s slide set evaluated at a time point, the mean of the raters scores for each subject will be formed.

For each person with PN that received selumetinib, the paired difference between baseline and pre-cycle 13 of these mean scores will be determined.

For the full set of approximately 35 paired scores, the difference will be assessed for statistical importance by means of a paired t-test, or a Wilcoxon signed rank test.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Clinician Raters - those who are professionally involved with direct patient care and have a career in the medical field and familiar with NF1 (Cohort 1A), OR

Clinician Raters - those who are professionally involved with direct patient care and have a career in the medical field but are not familiar with NF1 (Cohort 1B), OR

Non-clinician Raters - those who are not professionally involved in direct patient care or do not have a career in the medical field, but who are a first or second degree relative of a subject with NF1 or are otherwise closely associated with a subject with NF1 and familiar with NF1 (Cohort 2A), OR

Non-clinician Raters - those who are not professionally involved in direct patient care or do not have a career in the medical field, and who are not a first or second degree relative of a subject with NF1 and are otherwise not closely associated with a subject with NF1 (Cohort 2B)

* Age greater than or equal to18 years.
* The ability of a subject to understand and the willingness to sign a written informed consent document.
* Ability to read and write in English.

EXCLUSION CRITERIA:

* Raters should not be employees of the NIH.
* Raters should not be directly involved in the NCI Phase 1/2 study of selumetinib (11-C-0161), either as an investigator or as a subject or first-degree family member of a subject enrolled on the trial.

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Clinicians and non-clinician raters familiar with NF1; Participants enrolled on NIH protocols 11-C-0161 and 08-C-0079 with NF1 and visible plexiform neurofibromas
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the degree of changes in disfigurement measures | ongoing
  Mean scores for disfigurement as determined by raters reviewing photographs before treatment and just prior to cycle 13 of treatment.

SECONDARY OUTCOMES:
Differences in the disfigurement scores assigned by raters between cohorts of clinical raters who differ by NF1 familiarity and non-clinical raters who differ by NF1 familiarity | ongoing
  mean scores for disfigurement will be compared using a paired t-test or Wilcoxon signed rank test
Correlation between achieving a partial response on selumetinib and having an improvement in PN-related disfigurement | ongoing
  changes in score will be compared using a Wilcoxon rank sum test
Intra-reliability of a novel disfigurement scale among raters | ongoing
  scores for disfigurement at initial evaluation and a subsequent evaluation to assess reliability will be obtained and subtracted to form the difference in each score at the two time points
Correlation between the degree of change in disfigurement and percentage of PN volume shrinkage | ongoing
  Spearman correlation analysis to assess the degree of change in disfigurement and percentage of PN volume shrinkage from baseline
Factors most important in causing change in disfigurement | ongoing
  descriptive statistical analysis of factors
Agreement among raters within a cohort with respect to the evaluation of disfigurement to assess the reliability of a novel disfigurement scale | ongoing
  Full set of 15 pairwise Kappa statistics, taken two at a time will be constructed. For the full set of 15 Kappa statistics, the mean value along with a two-sided 95% confidence interval, will be reported separately for each of the 4 cohorts.
Feasibility of understanding and completing a novel disfigurement scale | ongoing
  descriptive findings of questionnaire responses
Overall difference among the 4 cohorts of raters with respect to scores assigned for disfigurement | ongoing
  mean scores for disfigurement will be compared using ANOVA or Kruskal-Wallis test as appropriate
PN-related disfigurement rating consistency with subject/parent responses to Global Impression of Change (GIC) | ongoing
  descriptive findings of ratings compared to Global Impression of Change (GIC) responses

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Gross, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
.All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Derived] John L, Singh G, Dombi E, Wolters PL, Martin S, Baldwin A, Steinberg SM, Bernstein J, Whitcomb P, Pichard DC, Dufek A, Gillespie A, Heisey K, Bornhorst M, Fisher MJ, Weiss BD, Kim A, Widemann BC, Gross AM. Development and pilot validation of a novel disfigurement severity scale for plexiform neurofibromas in children with neurofibromatosis type 1. Clin Trials. 2024 Apr;21(2):189-198. doi: 10.1177/17407745231206402. Epub 2023 Oct 25. PMID 37877369
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000173-C.html